CLINICAL TRIAL: NCT00476996
Title: A Randomized, Double-Blind, Parallel Group, International Study to Evaluate the Safety and Efficacy of Ocrelizumab Compared to Placebo in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to at Least One Anti-TNF-α Therapy
Brief Title: A Study of Ocrelizumab Compared to Placebo in Patients With Active Rheumatoid Arthritis Who Don't Have a Response to Anti-TNF-α Therapy (SCRIPT)
Acronym: SCRIPT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment was fully completed for this study; however, the study was terminated during conduct after the primary endpoint analysis was completed.
Sponsor: Genentech, Inc. (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT3986g; WA20495 (Other: Genentech); 2006-005330-20 (EudraCT Number)
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; SCRIPT; anti-CD20; CD20
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Leflunomide; Methotrexate; ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ocrelizumab 200 mg x 2 IV + Non-Biologic DMARD Therapy (Experimental): Participants will receive 2 intravenous (IV) infusions of 200 milligram (mg) of ocrelizumab, separated by 14 days (Day 1 and Day 15) in combination with any non-biologic DMARD
  Interventions: Drug: Leflunomide; Drug: Methotrexate; Drug: Ocrelizumab
- Ocrelizumab 500 mg x 2 IV + Non-Biologic DMARD Therapy (Experimental): Participants will receive 2 IV infusions of 500 mg of ocrelizumab, separated by 14 days (Day 1 and Day 15) in combination with any non-biologic DMARD
  Interventions: Drug: Leflunomide; Drug: Methotrexate; Drug: Ocrelizumab
- Placebo x 2 IV + Non-Biologic DMARD Therapy (Placebo Comparator): Participants will receive ocrelizumab matching placebo IV in two infusions, separated by 14 days (Day 1 and Day 15) in combination with any non-biologic DMARD
  Interventions: Drug: Leflunomide; Drug: Methotrexate; Drug: Placebo

INTERVENTIONS:
Drug: Leflunomide — Oral repeating dose
Drug: Methotrexate — Oral or parenteral repeating dose
Drug: Ocrelizumab — Intravenous repeating dose (200mg)
  Arms: Ocrelizumab 200 mg x 2 IV + Non-Biologic DMARD Therapy
Drug: Ocrelizumab — Intravenous repeating dose (500mg)
  Arms: Ocrelizumab 500 mg x 2 IV + Non-Biologic DMARD Therapy
Drug: Placebo — Intravenous repeating dose
  Arms: Placebo x 2 IV + Non-Biologic DMARD Therapy

SUMMARY:
This study will evaluate the efficacy and safety of ocrelizumab, compared with placebo, in patients with active rheumatoid arthritis who have an inadequate response to at least one anti-TNF-alpha therapy. Patients will be randomized to receive placebo, 200mg of intravenous ocrelizumab, or 500mg of i.v. ocrelizumab on days 1 and 15. A repeat course of i.v. treatment will be administered at weeks 24 and 26. All patients will receive stable doses of either concomitant methotrexate (7.5-25mg/week) or leflunomide (10-20mg po daily) and may receive additional DMARDs. The treatment period is planned for 48 weeks (until primary analysis) and then participants will enter the open label phase until the drug is commercialized. Target sample size is 1000.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ 18 years of age
* Rheumatoid arthritis for at least 3 months
* Inadequate response to previous or current treatment with at least one anti-TNF-alpha agent
* Receiving either leflunomide or methotrexate for ≥ 12 weeks, with a stable dose for the last 4 weeks
* Swollen joint count (SJC) ≥ 4 (66 joint count) and tender joint count (TJC) ≥ 4 (68 joint count) at screening and baseline.
* CRP ≥ 0.6 mg/dL using a high-sensitivity assay.
* Positive rheumatoid factor or positive anti-CCP antibody or both.

Exclusion Criteria:

* Rheumatic autoimmune disease or inflammatory joint disease, other than RA
* Any surgical procedure in past 12 weeks,or planned within 48 weeks of baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 836 (Actual)
Dates: Start 2007-05-15 (Actual); Primary Completion 2010-01-21 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (266):
- United States (144):
  - Pinnacle Research Group; Llc, Central, Anniston, Alabama
  - Rheumatology Associates, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, Huntsville, Alabama
  - Arizona Arthritis & Rheumatology Research, Pllc, Mesa, Arizona
  - Arthrocare, Arthritis Care and Research, P.C., Mesa, Arizona
  - Catalina Pointe Clinical Research, Inc., Tucson, Arizona
  - Uni of Arizona Health Science Center; Dept of Rheumatology/Immunology, Tucson, Arizona
  - CHI St. Vincent Medical Group Hot Springs, Hot Springs, Arkansas
  - Little Rock Diagnostic Clinic, Little Rock, Arkansas
  - Allergy & Rheumatology Centre, La Jolla, California
  - Private Practice, Long Beach, California
  - Valerius Medical Group & Research Ctr of Greater Long Beach, Los Alamitos, California
  - Uni of Southern California School of Medicine, Los Angeles, California
  - Pacific Arthritis Care Center, Los Angeles, California
  - Stanford Uni Medical Center; Divison of Rheumatology, Palo Alto, California
  - Ucsd, Dept of Medicine; Rheumatology, San Diego, California
  - San Diego Arthritis Med Clnc, San Diego, California
  - East Bay Rheumatology, San Leandro, California
  - Arthritis Treatment Center of South Bay, Torrance, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Arthritis Assoc & Osteoporosis; Ctr of Colorado Springs, Colorado Springs, Colorado
  - Arthritis & Osteoporosis Center P.C., Camden, Connecticut
  - New England Research Associates, Trumbull, Connecticut
  - Rheumatolgy Consultants of Deleware, Lewes, Delaware
  - Javed Rheumatology Associates, Inc., Newark, Delaware
  - Arthritis & Rheumatism; Disease Specialities, Aventura, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Arthritis Center Palm Harbor, Palm Harbor, Florida
  - Arthritis Rsrch of Florida, Inc., Palm Harbor, Florida
  - Sarasota Arthritis Center; Research Dept, Sarasota, Florida
  - Center For Arthritis; Research Dept, South Miami, Florida
  - SW Florida Clinical Research, Tampa, Florida
  - Tampa General Hospital; Rheumatology Research Dept, Tampa, Florida
  - Burnette & Silverfield, MDS, Tampa, Florida
  - Florida Medical Center, Zephyrhills, Florida
  - Atlanta Center For Clinical Research., Atlanta, Georgia
  - Csi Research, Inc., Cumming, Georgia
  - Marietta Rheumatology Associates, Pc, Marietta, Georgia
  - Intermountain Orthopaedics, Boise, Idaho
  - Coeur D'Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - Idaho Arthritis Center, Meridian, Idaho
  - Uni of Chicago, Chicago, Illinois
  - Evanston Northwestern Healthcare; Rheumatology, Evanston, Illinois
  - Quad City Rheumatology, Sc, Moline, Illinois
  - Illinois Bone & Joint Inst., Morton Grove, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Iu Outpatient Clinical Research Facility, Indianapolis, Indiana
  - Diagnostic Rheumatology & Research, Indianapolis, Indiana
  - Medical Specialists Clinical Research Center, Munster, Indiana
  - Physician'S Clinic of Iowa, Cedar Rapids, Iowa
  - Uni of Kansas Medical Center, Kansas City, Kansas
  - Center For Arthritis & Osteoporosis, Elizabethtown, Kentucky
  - Bluegrass Comm Research, Inc., Lexington, Kentucky
  - Kentuckiana Center For Better Bone & Joint Healthx, Louisville, Kentucky
  - Baton Rouge Clinic, Amc, Baton Rouge, Louisiana
  - Johns Hopkins University; Department of Rheumatology, Baltimore, Maryland
  - Center For Rheumatology & Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Clinsite;Research Division of Integrated Health Associates, Ann Arbor, Michigan
  - Rheumatology, P.C.; Medical Arts Building, Kalamazoo, Michigan
  - Borgess Research Institute, Kalamazoo, Michigan
  - Fiechtner Research Inc, Lansing, Michigan
  - Office of Andrew Sulich, Md, Saint Clair Shores, Michigan
  - St Luke's Whiteside Research, Duluth, Minnesota
  - St. Mary'S Duluth Clinic Health System; Rheumatology Dept, Duluth, Minnesota
  - St. Paul Rheumatology, Eagan, Minnesota
  - Park Nicollet Inst. ; Rtrc, Minneapolis, Minnesota
  - Jackson Arthritis Clinic, Flowood, Mississippi
  - North Mississippi Medical Ctr; Internal Medicine Associates, Tupelo, Mississippi
  - David S Rosenberg, Florissant, Missouri
  - St. John'S Health System Inc.; St. John'S Medical Research, Springfield, Missouri
  - Clayton Medical Research, St Louis, Missouri
  - Physicians Group, LC DBA Rheumatology & Internal Medicine Associates, St Louis, Missouri
  - Arthritis Consultants, St Louis, Missouri
  - Westroads Medical Group, Omaha, Nebraska
  - Seacoast Arthritis and Osteoporosis Center, Dover, New Hampshire
  - Nashua Rheumatology - Foundation Medical Partners, Nashua, New Hampshire
  - Mark Fisher Md, Facr, Llc, Haddon Heights, New Jersey
  - Arthritis Rheumatic & Back Disease Associates, Voorhees Township, New Jersey
  - The Center of Rheumatology, Albany, New York
  - Arthritis & Osteoporosis Center, Brooklyn, New York
  - Southern Tier Arthritis & Rheumatism, Olean, New York
  - Aair Research Center, Rochester, New York
  - Andrew Porges Pc, Roslyn, New York
  - Rheumatology Associates of Long Island, Smithtown, New York
  - Asheville Arthritis & Osteoporosis Center, PA, Asheville, North Carolina
  - Arthritis Associates, Belmont, North Carolina
  - Metrolina Medical Research, Charlotte, North Carolina
  - Carolina Bone & Joint P.A., Charlotte, North Carolina
  - Physicians East Pa, Greenville, North Carolina
  - St. Alexius Medical Center; Arthritis Clinic, Bismarck, North Dakota
  - Deaconess Arthritis Center; Rheumatic Disease Study Group, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Stat Research, Inc, Dayton, Ohio
  - David Mandel Inc, Mayfield, Ohio
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Health Research of Oklahoma, Llc, Oklahoma City, Oklahoma
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Oklahoma Center For Arthritis Therapy & Research, Tulsa, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Pro Research, Eugene, Oregon
  - Portland Rheumatology Clinic Llc, Lake Oswego, Oregon
  - Providence Arthritis Center, Portland, Oregon
  - East Penn Rheumatology Associates, Pc, Bethlehem, Pennsylvania
  - Arthritis Associates, Erie, Pennsylvania
  - Rheumatology Associates of NW Pa, Erie, Pennsylvania
  - Arthritis Group, Philadelphia, Pennsylvania
  - Advanced Rheumatology & Arthritis Research Center, Wexford, Pennsylvania
  - Clinical Research Center of Reading, Wyomissing, Pennsylvania
  - Low Country Research Center, Charleston, South Carolina
  - Palmetto Clinical Trial Services, LLC, Fountain Inn, South Carolina
  - Unifour Medical Research Associates, Hickory Grove, South Carolina
  - Medical Uni of South Carolina, North Charleston, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Rheumatology Consultants, Knoxville, Tennessee
  - Arthritis Group, Memphis, Tennessee
  - Ramesh Gupta - PP, Memphis, Tennessee
  - Aamr Research Clinic, Amarillo, Texas
  - Amarillo Center For Clinical Research, Amarillo, Texas
  - Austin Rheumatology Research, Austin, Texas
  - Walter F. Chase, Md, Pa, Austin, Texas
  - Arthritis Care & Diagnostic Center, Dallas, Texas
  - Arthritis Care and Research Centre, Dallas, Texas
  - Metroplex Clinical Research, Dallas, Texas
  - Arthritis Centers of Texas, Dallas, Texas
  - Uni of Texas Southwestern Medical Center; Internal Medicine, Dallas, Texas
  - Arthritis & Osteoporosis Associates, LLP, Lubbock, Texas
  - Southwest Rheumatology, Mesquite, Texas
  - Radiant Research, San Antonio, Texas
  - Texas Arthritis Research Center; Center for Arthritis & Rheumatic Diseases, San Antonio, Texas
  - Texas Research Center, Sugar Land, Texas
  - Uni of Utah Medical Center, Salt Lake City, Utah
  - Arthritis Clinic of Northern Virginia, Arlington, Virginia
  - Sentara Medical Group, Norfolk, Virginia
  - Seattle Rheumatology Associates, Seattle, Washington
  - Arthritis Northwest, Spokane, Spokane, Washington
  - Office of George Krick, Md, Tacoma, Washington
  - Tacoma Center For Arthritis Research, Tacoma, Washington
  - Vancouver Clinic; Research Dept, Vancouver, Washington
  - Clinical Trials Northwest, Yakima, Washington
  - Rheumatic Disease Center, Glendale, Wisconsin
  - Gundersen Clinic Ltd;Sec. Rheumatology/Dept. of Internal Med, Onalaska, Wisconsin
- Argentina (3):
  - Organizacion Medica de Investigacion, Buenos Aires
  - Inst. de Rehabilitacion Psicofisica; Reumathology, Buenos Aires
  - CER Instituto Médico; REUMATOLOGÍA, San Juan Bautista
- Australia (3):
  - Sunshine Coast Rheumatology Research Unit, Maroochydore, Queensland
  - Princess Alexandra Hospital; Rheumatology, Woolloongabba, Queensland
  - Royal Perth Hospital; Rheumatology, Shenton Park, Western Australia
- Belgium (7):
  - AZ Sint Jan, Bruges
  - CHU Brugmann (Victor Horta), Brussels
  - CHU de Charleroi, Charleroi
  - UZ Gent, Ghent
  - GHdC Site Saint-Joseph, Gilly (Charleroi)
  - UZ Leuven Gasthuisberg, Leuven
  - ZNA Jan Palfijn, Merksem
- Brazil (5):
  - Centro Internacional de Pesquisa; Reumatologia, Goiânia, Goiás
  - Centro de Estudos em Terapias Inovadoras - CETI, Curtiba, Paraná
  - Hospital Universitario Clementino Fraga Filho - UFRJ; Reumatologia, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clinicas - UNICAMP, Campinas, São Paulo
  - Hospital Abreu Sodre - AACD;Pesquisa Clinica, São Paulo, São Paulo
- Canada (16):
  - The Governors of the Uni of Alberta; Heritage Medical Research Centre, Edmonton, Alberta
  - Arthritis Research Centre, Vancouver, British Columbia
  - Manitoba Clinic, Winnipeg, Manitoba
  - Wharton Medical Clinic; Burlington, Burlington, Ontario
  - Mac Research Inc., Hamilton, Ontario
  - K-W Musculoskeletal Research, Kitchener, Ontario
  - St. Joseph'S Health Care Centre; Rheumatology, London, Ontario
  - Credit Valley, Rheumatology, Mississauga, Ontario
  - The Ottawa Hospital - Riverside Campus; the Arthritis Centre, Ottawa, Ontario
  - University Health Network; Toronto Western Hospital, Toronto, Ontario
  - Hopital Maisonneuve- Rosemont; Rheumatology, Montreal, Quebec
  - Institut de Rhumatologie de Montreal, Montreal, Quebec
  - Montreal Rheumatic Disease Centre, Montreal, Quebec
  - Groupe de Recherche En Rhumatologie Et Maladies Osseuses, Québec, Quebec
  - Clin. de Rhumatologie, Trois-Rivières, Quebec
  - Royal Uni Hospital; Medicine Dept, Saskatoon, Saskatchewan
- Revmatologicky Ustav, Prague, Czechia
- France (10):
  - Hopital De Bois Guillaume; Rhumatologie, Bois-Guillaume
  - CH Jean Rougier; Rhumato Reed Fonctionnelle, Cahors
  - Hopital Louis Pasteur; Service De Medecine Interne et de Rhumatologie, Colmar
  - CH Du Mans; Rhumatologie, Le Mans
  - Hopital B Roger Salengro; Rhumatologie, Lille
  - Fondation Hopital Saint Joseph; Rhumatologie, Marseille
  - Hopital Lapeyronie; Immunologie Rhumatologie, Montpellier
  - Hopital de L'Archet; Rhumatologie, Nice
  - Hopital Cochin; Rhumatologie A, Paris
  - Hopital Cochin; Rhumatologie B, Paris
- Germany (16):
  - Praxis Dr. med. Reiner Kurthen, Aachen
  - Schlosspark Klinik; Abt. Rheumatologie, Berlin
  - Klinik der Uni zu Köln; Klinik für Innere Medizin, Cologne
  - Klinik Duisburg; Klinik Für Rheumatologie, Duisburg
  - Endokrinologikum Frankfurt; Rheumatologie & Gynäkologie, Frankfurt
  - Universitätsklinikum Freiburg; Medizinische UNI-Klinik; Abt. Innere Medizin - VI Rheumatologie, Freiburg im Breisgau
  - Internistisches Praxiszentrum Am Krankenhaus Balserische Stiftung; Innere Medizin / Rheumatologie, Giessen
  - Evangelisches Krankenhaus Hagen-Haspe Rheumaklinik, Hagen
  - Medizinische Hochschule Zentrum Innere Medizin Abt.Klinische Immunologie und Rheumatologie, Hanover
  - Rheumapraxis PD Dr.med. Bernhard Heilig, Heidelberg
  - UNI-Klinikum Heidelberg Medizinische Klinik Innere Medizin V, Heidelberg
  - Fachärzte für Innere Medizin - Rheumatologie - Dr. med. Ino Gao und Dr. med. Maria Anna Meier, Heidelberg
  - Uniklinik Mainz; I. Medizinische Klinik, Mainz
  - Klinikum der Universitat Munchen; Bereich Pettenkoferstr; Rheumaeinheit der medizinischen Klinik IV, München
  - Rheumapraxis an der Hase, Osnabrück
  - Universitätsklinikum Würzburg; Medizinische Klinik und Poliklinik II; Hämatologie / Onkologie, Würzburg
- Hungary (4):
  - Orszagos Reumatologiai Es Fizioterapias Intezet, Budapest
  - Budai Irgalmasrendi Kórház KHT. II. Reumatológia, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum; Belgyógyászati Intézet, Reumatológiai Tanszék, Debrecen
  - Vas Megye Es Szombathely M.J.V. Markusovszky Korhaza, Szombathely
- Israel (5):
  - Assaf Harofe; Dept of Medicine B, Beer Yaakov
  - Soroka Medical Center; Reumatology, Beersheba
  - Meir Medical Center; Heamatology Dept, Kfar Saba
  - Beilinson Medical Center; Rheumatology, Petah Tikva
  - Sourasky / Ichilov Hospital; Rheumatology, Tel Aviv
- Italy (4):
  - Arcispedale Santa Maria Nuova; Reumatologia, Reggio Emilia, Emilia-Romagna
  - Università Degli Studi Di Genova - Dimi; Reumatologia, Genoa, Liguria
  - Irccs Policlinico San Matteo; Reumatologia Adulti, Pavia, Lombardy
  - Az. Osp. Pisana Ospedale S. Chiara; U.O. Di Reumatologia, Pisa, Tuscany
- Japan (14):
  - Seihoku Chuoh Hospital; Department Of Rheumatology, Aomori
  - Univ. of Occupational and Environmental Health; Rheumatology, Clinical Immunology and Medicine, Fukuoka
  - National Hospital Organization Kyushu Medical Center; Rheumatology and Internal Medicine, Fukuoka
  - Higashihiroshima Memorial Hospital; Rheumatology, Internal Medicine, Hiroshima
  - Hokkaido Uni Hospital; Second Department of Internal Medicine, Hokkaido
  - Matsubara Mayflower Hospital; Rheumatology, Hyōgo
  - Sasebo Chuo Hospital ; Internal Medicine, Nagasaki
  - Osaka Minami Medical Center; Rheumatoid Arthritis, Osaka
  - Saitama Medical University Hospital ; Rheumatology and Applied Immunology, Saitama
  - Saitama Medical Center/School; Rheumatology, Clinical immunology, Saitama
  - Seirei Hamamatsu General Hospital; Rheumatology, Shizuoka
  - Jichi Medical School Hospital; Rheumatology and Clinical Immunology, Tochigi
  - Tokyo Medical & Dental University; Medicine & Rheumatology, Tokyo
  - Tokyo Women's Medical University, Tokyo
- Mexico (4):
  - Consultorio Privado Dr. Javier Orozco, Guadalajara
  - Unidad de Reumatologia Rehabilitacion Integral; Centro Medico Del Angel, Mexicali
  - Unidad De Enfermedades; Cronico Degenerativas, SC., México
  - Clinica San Jose Obregon; Rheumatology, Obregón
- Netherlands (2):
  - Academisch Medisch Centrum; Division of Clinical Immunology & Rheumatology, Amsterdam
  - Maxima Medisch Centrum; Rheumatology, Eindhoven
- Timaru Hospital, Timaru, New Zealand
- Centro de Infusion Marbella; Consultorios Royal Center Num 214, Panama City, Panama
- Peru (3):
  - Hospital Alberto Sabogal Sologuren; Remautology, Callao
  - Clinica San Felipe; Consultorio de Reumatología, Lima
  - Hospital Nacional Edgardo Rebagliati Martins; Servicio de Reumatología, Lima
- Poland (3):
  - Szpital Uniwersytecki; nr 2 im. Dr J. Biziela, Bydgoszcz
  - Wojewodzki Szpital Zespolony; Oddzial Reumatologii, Elblag
  - Klinika Reumatologii I Chorób Wewn. Pum W Szczecinie; Samodzielny Publiczny Szpital Kliniczny Nr 1, Szczecin
- Narodny Ustav Reumatickych Chorob - 34479; Rheumatology, Piešťany, Slovakia
- Bolnica dr. Petra Drzaja, Klinicni center Ljubljana; Klinicni oddelek za revmatologijo, Ljubljana, Slovenia
- Spain (13):
  - Corporacio Sanitaria Parc Tauli; Servicio de Reumatologia, Sabadell, Barcelona
  - Hospital de Jerez de la Frontera; Servicio de Reumatologia, Jerez de la Frontera, Cadiz
  - Hospital Sierrallana; Servicio de Reumatologia, Torrelavega, Cantabria
  - Complejo Hospitalario Universitario A Coruña (CHUAC); Servicio de Reumatologia, A Coruña, LA Coruña
  - Hospital Univ. Central de Asturias; Servicio de Reumatologia, Oviedo, Principality of Asturias
  - Hospital de Basurto; Servicio de Reumatologia, Bilbao, Vizcaya
  - Hospital Universitario Infanta Cristina; Servicio de Reumatologia, Badajoz
  - Hospital Clinic i Provincial; Servicio de Reumatologia, Barcelona
  - Hospital Universitari de Bellvitge; Servicio de Reumatologia, Barcelona
  - Complejo Asistencial Universitario de Burgos; Servicio de Reumatología, Burgos
  - Hospital General Universitario de Guadalajara; Servicio de Reumatologia, Guadalajara
  - Hospital Universitario 12 de Octubre; Servicio de Reumatologia, Madrid
  - Hospital Clinico Universitario de Salamanca; Servicio de Reumatologia, Salamanca
- Sweden (2):
  - Uni Hospital Linkoeping; Dept. of Rheumatology, Linköping
  - Akademiska sjukhuset, Reumatologkliniken, Uppsala
- Switzerland (2):
  - CHUV; Hôpital orthopédique, Rhumatologie, Lausanne
  - Universitätsspital Zürich; Klinik für Rheumatologie, Zurich
- Chang Gung Medical Foundation - Kaohsiung; Rheumatology, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Emery P, Rigby W, Tak PP, Dorner T, Olech E, Martin C, Millar L, Travers H, Fisheleva E. Safety with ocrelizumab in rheumatoid arthritis: results from the ocrelizumab phase III program. PLoS One. 2014 Feb 3;9(2):e87379. doi: 10.1371/journal.pone.0087379. eCollection 2014. PMID 24498318
- [Derived] Tak PP, Mease PJ, Genovese MC, Kremer J, Haraoui B, Tanaka Y, Bingham CO 3rd, Ashrafzadeh A, Travers H, Safa-Leathers S, Kumar S, Dummer W. Safety and efficacy of ocrelizumab in patients with rheumatoid arthritis and an inadequate response to at least one tumor necrosis factor inhibitor: results of a forty-eight-week randomized, double-blind, placebo-controlled, parallel-group phase III trial. Arthritis Rheum. 2012 Feb;64(2):360-70. doi: 10.1002/art.33353. PMID 22389919

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited across 25 countries.
Pre-assignment Details: The study population comprised of adult participants with active RA of >/= 3 months duration who had an inadequate clinical response due to toxicity or inadequate efficacy to previous or current treatment with one or more anti-TNF-alpha therapies.
Groups:
- Placebo x 2 IV + Non-Biologic DMARD: Participants received Ocrelizumab matching placebo intravenously (IV) in two infusions, separated by 14 days (Day 1 and Day 15) in combination with any non-biologic DMARD
- Ocrelizumab 200 mg x 2 + Non-Biologic DMARD: Participants received 2 intravenous (IV) infusions of 200 milligram (mg) of ocrelizumab (total 400 mg), separated by 14 days (Day 1 and Day 15) in combination with any non-biologic DMARD
- Ocrelizumab 500 mg x 2 + Non-Biologic DMARD: Participants received 2 intravenous (IV) infusions of 500 milligram (mg) of ocrelizumab (total 1000 mg), separated by 14 days (Day 1 and Day 15) in combination with any non-biologic DMARD
- Ocrelizumab 500 mg x 2 IV + Non-biologic DMARD (OLE): At the discretion of the investigator, eligible participants received 500 mg Ocrelizumab IV in two infusions separated by 14 days
Period: Blinded Treatment Phase (up to Week 48)
Arm/Group | Placebo x 2 IV + Non-Biologic DMARD | Ocrelizumab 200 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 IV + Non-biologic DMARD (OLE)
Started | 277 | 277 | 282 | 0
Completed | 205 | 222 | 237 | 0
Not Completed | 72 | 55 | 45 | 0
Not completed — Withdrawal by Subject | 12 | 7 | 7 | 0
Not completed — Protocol Violation | 1 | 3 | 0 | 0
Not completed — Early termination of the study | 24 | 20 | 21 | 0
Not completed — Non-Compliance with Study Drug | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 4 | 3 | 0
Not completed — Lack of Efficacy | 22 | 5 | 6 | 0
Not completed — Death | 2 | 1 | 1 | 0
Not completed — Adverse Event | 11 | 13 | 7 | 0
Period: OLE Phase (From Week 48)
Arm/Group | Placebo x 2 IV + Non-Biologic DMARD | Ocrelizumab 200 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 IV + Non-biologic DMARD (OLE)
Started | 0 | 0 | 0 | 664
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 664
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 50
Not completed — Adverse Event | 0 | 0 | 0 | 8
Not completed — Death | 0 | 0 | 0 | 7
Not completed — Lack of Efficacy | 0 | 0 | 0 | 13
Not completed — Lost to Follow-up | 0 | 0 | 0 | 4
Not completed — Non-Compliance with Study Drug | 0 | 0 | 0 | 4
Not completed — Early termination of the study | 0 | 0 | 0 | 578

BASELINE CHARACTERISTICS:
Population: Intent-toTreat (ITT) All randomized participants who received any part of an infusion of study medication were included in the ITT analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo x 2 IV + Non-Biologic DMARD | Ocrelizumab 200 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 + Non-Biologic DMARD | Total
Number analyzed (Participants) | 277 | 277 | 282 | 836
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (11.3) | 54.5 (11.2) | 53.8 (11.6) | 54.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215 | 214 | 236 | 665
  Male | 62 | 63 | 46 | 171
Race/Ethnicity, Customized [Number; unit: Participants]
  American indian or Alaska native | 9 | 8 | 9 | 26
  Asian (Indian Subcontinent) | 1 | 0 | 0 | 1
  Asian (Other than Indian subcontinent) | 39 | 38 | 38 | 115
  Black | 16 | 18 | 12 | 46
  Native Hawaiian or other Pacific Islander | 0 | 1 | 2 | 3
  Other | 6 | 11 | 14 | 31
  White | 206 | 201 | 207 | 614

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology 20 (ACR20) Responses
Description: ACR20 response: greater than or equal to (≥) 20% improvement in tender or swollen joint counts and 20% improvement in 3 of the following 5 criteria: 1) Physician's global assessment of disease activity, 2) participant assessment of disease activity, 3) Patient Assessment of Pain (visual analog scale [VAS]), 4) participant assessment of functional disability via a Health Assessment Questionnaire (HAQ), and 5) erythrocyte sedimentation rate (ESR) at each visit.
Time Frame: Weeks 24 and 48
Population: Intent-to-Treat (ITT) All randomized participants who received any part of an infusion of study medication were included in the ITT analysis. Number of participants for whom data were collected is indicated for each time point.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo x 2 IV + Non-Biologic DMARD | Ocrelizumab 200 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 + Non-Biologic DMARD
Number analyzed (Participants) | 277 | 277 | 282
Percentage
  Percentage of Responders at Week 24 | 22 [17.1 to 26.9] | 42.2 [36.4 to 48.1] | 47.9 [42.0 to 53.7]
  Percentage of Responders at Week 48 | 19.5 [14.8 to 24.2] | 48.7 [42.9 to 54.6] | 50.7 [44.9 to 56.5]
Statistical Analysis 1: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; At Week 24, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 20.4, 95% CI 2-sided [12.8 to 27.9]
Statistical Analysis 2: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; At Week 24, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 25.2, 95% CI 2-sided [17.7 to 32.7]
Statistical Analysis 3: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; At Week 48, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 29.1, 95% CI 2-sided [21.6 to 36.6]
Statistical Analysis 4: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; At Week 48, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 30.3, 95% CI 2-sided [22.8 to 37.7]

2. Secondary Outcome: Percentage of Participants With a Major Clinical Response
Description: Major clinical response was defined as achieving an ACR70 response and maintaining this response for a consecutive period of at least 6 months.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo x 2 IV + Non-Biologic DMARD | Ocrelizumab 200 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 + Non-Biologic DMARD
Number analyzed (Participants) | 277 | 277 | 282
Percentage | 1.8 [0.2 to 3.4] | 4.0 [1.7 to 6.3] | 5.7 [3.0 to 8.4]
Statistical Analysis 1: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; Analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p = 0.1885, Cochran-Mantel-Haenszel; Weighted Difference = 2.1, 95% CI 2-sided [-1.0 to 5.2]
Statistical Analysis 2: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; Analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p = 0.0330, Cochran-Mantel-Haenszel; Weighted Difference = 3.6, 95% CI 2-sided [0.3 to 6.8]

3. Secondary Outcome: Percentage of Participants Achieving Disease Activity Score (DAS28) Remission
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. DAS28 Remission is defined as a DAS28 score < 2.6.
Time Frame: Weeks 24 and 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo x 2 IV + Non-Biologic DMARD | Ocrelizumab 200 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 + Non-Biologic DMARD
Number analyzed (Participants) | 277 | 277 | 282
Percentage
  Percentage of Participants at Week 24 | 1.8 [0.2 to 3.4] | 5.8 [3.0 to 8.5] | 6.0 [3.3 to 8.8]
  Percentage of Participants at Week 48 | 1.4 [0.0 to 2.8] | 11.9 [8.1 to 15.7] | 12.1 [8.3 to 15.9]
Statistical Analysis 1: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; At Week 24, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p = 0.0175, Cochran-Mantel-Haenszel; Weighted Difference = 4.2, 95% CI 2-sided [0.7 to 7.6]
Statistical Analysis 2: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; At Week 24, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p = 0.0134, Cochran-Mantel-Haenszel; Weighted Difference = 4.3, 95% CI 2-sided [0.9 to 7.8]
Statistical Analysis 3: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; At Week 48, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 10.5, 95% CI 2-sided [6.2 to 14.8]
Statistical Analysis 4: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; At Week 48, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 10.5, 95% CI 2-sided [6.2 to 14.7]

4. Secondary Outcome: Change in DAS28 From Baseline
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10.
Time Frame: Weeks 24 and 48
Population: Intent-to-Treat (ITT) All randomized participants who received any part of an infusion of study medication were included in the ITT analysis Number of participants for whom data were collected is indicated for each time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo x 2 IV + Non-Biologic DMARD | Ocrelizumab 200 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 + Non-Biologic DMARD
Number analyzed (Participants) | 277 | 277 | 282
Score on a scale
  Baseline | 6.50 (1.014) | 6.47 (1.217) | 6.44 (1.039)
  Week 24: number analyzed (Participants) | 173 | 233 | 228
  Week 24 | -0.99 (1.166) | -1.60 (1.307) | -1.91 (1.349)
  Week 48: number analyzed (Participants) | 135 | 208 | 209
  Week 48 | -1.13 (1.404) | -2.11 (1.348) | -2.38 (1.496)
Statistical Analysis 1: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; Week 24 analysis using adjusted mean difference. Model contains region, baseline DMARD therapy, baseline DAS28 score and treatment; Test type: Superiority; p < 0.0001, Analysis of Variance; Adjusted Mean Difference = -0.6, 95% CI 2-sided [-0.8 to -0.3]
Statistical Analysis 2: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Analysis of Variance; Adjusted Mean Difference = -0.9, 95% CI 2-sided [-1.1 to -0.6]
Statistical Analysis 3: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; Week 48 analysis using adjusted mean difference. Model contains region, baseline DMARD therapy, baseline DAS28 score and treatment; Test type: Superiority; p < 0.0001, Analysis of Variance; Adjusted Mean Difference = -0.9, 95% CI 2-sided [-1.2 to -0.7]
Statistical Analysis 4: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p < 0.0001, Analysis of Variance; Adjusted Mean Difference = -1.2, 95% CI 2-sided [-1.5 to -0.9]

5. Secondary Outcome: Percentage of Participants With EULAR Response Rates of Good/ Moderate
Description: The EULAR response rate was based on the assessment of disease activity using the DAS28. The EULAR response criteria included not only change in disease activity but current disease activity. To be classified as responders, participants had to have a significant change in DAS28 and a low current disease activity. There were 4 categories of EULAR response rates: good, moderate, good/moderate, and none.
Time Frame: Weeks 24 and 48
Population: as for outcome 1
Measure: Number; unit: Percentage
Arm/Group | Placebo x 2 IV + Non-Biologic DMARD | Ocrelizumab 200 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 + Non-Biologic DMARD
Number analyzed (Participants) | 277 | 277 | 282
Percentage
  Week 24 | 31.4 | 54.2 | 61.0
  Week 48 | 24.9 | 58.8 | 60.3
Statistical Analysis 1: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; At Week 24, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Proportional Odds Analysis; Odds Ratio (OR) = 2.60, 95% CI 2-sided [1.85 to 3.66]
Statistical Analysis 2: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; At Week 24, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Proportional Odds Analysis; Odds Ratio (OR) = 3.49, 95% CI 2-sided [2.49 to 4.91]
Statistical Analysis 3: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; At Week 48, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Proportional Odds Analysis; Odds Ratio (OR) = 4.18, 95% CI 2-sided [2.93 to 5.96]
Statistical Analysis 4: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; At Week 48, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Proportional Odds Analysis; Odds Ratio (OR) = 5.04, 95% CI 2-sided [3.54 to 7.18]

6. Secondary Outcome: Percentage of Participants Achieving an ACR50 Response
Description: ACR50 response is defined as a ≥ 50% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: physician's global assessment of disease activity (MDG), patient's global assessment of disease activity (PGA), patient's assessment of pain, Health Assessment Questionnaire with Disability Index (HAQ-DI), and C-Reactive Protein (CRP).
Time Frame: Weeks 24 and 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo x 2 IV + Non-Biologic DMARD | Ocrelizumab 200 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 + Non-Biologic DMARD
Number analyzed (Participants) | 277 | 277 | 282
Percentage
  Percentage of Participants at Week 24 | 7.9 [4.8 to 11.1] | 21.3 [16.5 to 26.1] | 24.8 [19.8 to 29.9]
  Percentage of Participants at Week 48 | 9 [5.7 to 12.4] | 28.5 [23.2 to 33.8] | 30.9 [25.5 to 36.2]
Statistical Analysis 1: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; At Week 24, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 13.2, 95% CI 2-sided [7.4 to 19.1]
Statistical Analysis 2: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; At Week 24, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 16.2, 95% CI 2-sided [10.2 to 22.1]
Statistical Analysis 3: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; At Week 48, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 19.3, 95% CI 2-sided [12.9 to 25.6]
Statistical Analysis 4: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; At Week 48, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 20.8, 95% CI 2-sided [14.5 to 27.1]

7. Secondary Outcome: Percentage of Participants Achieving an ACR70 Response
Description: ACR70 response is defined as a ≥ 70% improvement (reduction) compared with Baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: physician's global assessment of disease activity (MDG), patient's global assessment of disease activity (PGA), patient's assessment of pain, HAQ-DI and CRP.
Time Frame: Weeks 24 and 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo x 2 IV + Non-Biologic DMARD | Ocrelizumab 200 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 + Non-Biologic DMARD
Number analyzed (Participants) | 277 | 277 | 282
Percentage
  Percentage of Participants at Week 24 | 2.9 [0.9 to 4.9] | 7.6 [4.5 to 10.7] | 9.9 [6.4 to 13.4]
  Percentage of Participants at Week 48 | 4.3 [1.9 to 6.7] | 11.2 [7.5 to 14.9] | 18.1 [13.6 to 22.6]
Statistical Analysis 1: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; At Week 24, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p = 0.0203, Cochran-Mantel-Haenszel; Weighted Difference = 4.6, 95% CI 2-sided [0.7 to 8.5]
Statistical Analysis 2: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; At Week 24, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p = 0.0014, Cochran-Mantel-Haenszel; Weighted Difference = 6.7, 95% CI 2-sided [2.6 to 10.8]
Statistical Analysis 3: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; At Week 48, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p = 0.0042, Cochran-Mantel-Haenszel; Weighted Difference = 6.6, 95% CI 2-sided [2.1 to 11.2]
Statistical Analysis 4: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; At Week 48, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 13.4, 95% CI 2-sided [8.2 to 18.6]

8. Secondary Outcome: Percentage of Participants With a Reduction in the HAQ-DI Score
Description: Health Assessment Questionnaire - Disability Index (HAQ-DI): The Stanford Health Assessment Questionnaire disability index is a patient reported questionnaire specific for RA. It consists of 20 questions referring to eight component. Reduction in the HAQ-DI score of 0.25 units from baseline to weeks 24 and 48 represented a minimal clinically relevant improvement.
Time Frame: Weeks 24 and 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo x 2 IV + Non-Biologic DMARD | Ocrelizumab 200 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 + Non-Biologic DMARD
Number analyzed (Participants) | 277 | 277 | 282
Percentage
  Percentage of Participants at Week 24 | 32.9 [27.3 to 38.4] | 52.3 [46.5 to 58.2] | 58.5 [52.8 to 64.3]
  Percentage of Participants at Week 48 | 23.1 [18.1 to 28.1] | 50.5 [44.7 to 56.4] | 51.8 [45.9 to 57.6]
Statistical Analysis 1: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; At Week 24, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 19.4, 95% CI 2-sided [11.3 to 27.5]
Statistical Analysis 2: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; At Week 24, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 24.7, 95% CI 2-sided [16.8 to 32.7]
Statistical Analysis 3: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 200 mg x 2 + Non-Biologic DMARD; At Week 48, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 27.2, 95% CI 2-sided [19.5 to 34.9]
Statistical Analysis 4: Comparison: Placebo x 2 IV + Non-Biologic DMARD vs Ocrelizumab 500 mg x 2 + Non-Biologic DMARD; At Week 48, analysis was stratified by region and baseline DMARD therapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Weighted Difference = 27.6, 95% CI 2-sided [20.0 to 35.3]

ADVERSE EVENTS:
Time Frame: From Day 1 to Week 48 and Week 96
Description: The safety population included all participants who received at least one treatment with study medication. In the safety population patients are categorized as treated, the ITT population as randomized. One patient randomized to Placebo and one patient randomized to the OCR 200 mg group, received at least one dose of OCR 500 mg.
Arm/Group | Placebo x 2 IV + Non-Biologic DMARD | Ocrelizumab 200 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 + Non-Biologic DMARD | Ocrelizumab 500 mg x 2 IV + Non-biologic DMARD (OLE)
All-Cause Mortality (participants affected / at risk) | 5/276 | 2/276 | 4/284 | 11/664
Serious Adverse Events (participants affected / at risk) | 41/276 | 46/276 | 40/284 | 138/664
Other Adverse Events (participants affected / at risk) | 152/276 | 153/276 | 158/284 | 361/664
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo x 2 IV + Non-Biologic DMARD (N=276) | Ocrelizumab 200 mg x 2 + Non-Biologic DMARD (N=276) | Ocrelizumab 500 mg x 2 + Non-Biologic DMARD (N=284) | Ocrelizumab 500 mg x 2 IV + Non-biologic DMARD (OLE) (N=664)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 2 | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 2
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 2 | 1 | 6
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Basedow's disease (Endocrine disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 4
Death (General disorders) | 0 | 0 | 1 | 1
Device dislocation (General disorders) | 0 | 0 | 0 | 1
Lead dislodgement (General disorders) | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2
Sudden death (General disorders) | 0 | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1
Surgical failure (General disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 1 | 1
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Bronchitis pneumococcal (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1
Bursitis infective (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 3 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 2
Escherichia pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Extradural abscess (Infections and infestations) | 0 | 0 | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 2
Genitourinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Implant site infection (Infections and infestations) | 1 | 0 | 0 | 0
Incision site cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Infectious colitis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 5 | 1 | 11
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 2 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 2 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Sycosis barbae (Infections and infestations) | 0 | 0 | 1 | 0
Serratia infection (Infections and infestations) | 1 | 0 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 2
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteochondroitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 7 | 4 | 4 | 7
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Wrist deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 2
Radiculitis lumbosacral (Nervous system disorders) | 0 | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 3
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 2
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 2
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Pleura effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0/275 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Physical assault (Social circumstances) | 0 | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1
Hernia repair (Surgical and medical procedures) | 0 | 1 | 0 | 0
Arteritis (Vascular disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2 | 3
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 1 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo x 2 IV + Non-Biologic DMARD (N=276) | Ocrelizumab 200 mg x 2 + Non-Biologic DMARD (N=276) | Ocrelizumab 500 mg x 2 + Non-Biologic DMARD (N=284) | Ocrelizumab 500 mg x 2 IV + Non-biologic DMARD (OLE) (N=664)
Darrhoea (Gastrointestinal disorders) | 10 | 15 | 15 | 0
Nausea (Gastrointestinal disorders) | 15 | 11 | 10 | 0
Bronchitis (Infections and infestations) | 19 | 28 | 22 | 64
Influenza (Infections and infestations) | 9 | 7 | 15 | 0
Nasopharyngitis (Infections and infestations) | 31 | 28 | 22 | 69
Sinusitis (Infections and infestations) | 14 | 13 | 13 | 53
Upper respiratory tract infection (Infections and infestations) | 36 | 37 | 45 | 96
Urinary tract infection (Infections and infestations) | 23 | 19 | 24 | 78
Infusion related reaction (Injury, poisoning and procedural complications) | 25 | 41 | 41 | 128
Headache (Nervous system disorders) | 15 | 12 | 15 | 0
Insomnia (Psychiatric disorders) | 12 | 9 | 16 | 0
Hypertension (Vascular disorders) | 21 | 18 | 19 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.